CLINICAL TRIAL: NCT00366379
Title: An Open Label Study to Determine the Effect on Fasting Glucose Levels, and Safety, of Increasing Doses of GK Activator (2) in Patients With Type 2 Diabetes Not Optimally Controlled With One Previous Oral Antihyperglycemic Agent.
Brief Title: A Dose-Titration Study of GK Activator (2) in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC19800
Record Dates: First submitted 2006-08-16; First posted 2006-08-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2)
- 2 (Experimental)
  Interventions: Drug: GK Activator (2)
- 3 (Experimental)
  Interventions: Drug: GK Activator (2)
- 4 (Experimental)
  Interventions: Drug: GK Activator (2)
- 5 (Experimental)
  Interventions: Drug: GK Activator (2)

INTERVENTIONS:
Drug: GK Activator (2) — 25-200mg po bid for 20 weeks

SUMMARY:
This study will assess the efficacy, safety and tolerability of increasing doses of GK Activator (2) in patients with type 2 diabetes whose condition has not been optimally controlled with one previous oral antihyperglycemic agent. After a 2 week washout from their previous antidiabetic therapy, patients will receive GK Activator (2) orally, twice a day for 12 weeks, at increasing doses of 25mg bid to 200mg bid; doses will be titrated to achieve a target fasting glucose level (FPG) of <100mg/dL. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes mellitus treated with one oral antihyperglycemic agent for >=3 months prior to screening.

Exclusion Criteria:

* type 1 diabetes mellitus;
* treatment with insulin, PPAR agonists or systemic corticosteroids during the 3 months prior to screening;
* women who are pregnant, breast-feeding or not using adequate contraceptive methods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients at each dose who achieve FPG <100mg/dL. | Throughout study

SECONDARY OUTCOMES:
Mean change in HbA1c and FPG from baseline to endpoint; absolute/relative changes in lipid profile. | At intervals throughout study
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (10):
  - Chandler, Arizona
  - Oviedo, Florida
  - Nampa, Idaho
  - Evansville, Indiana
  - Butte, Montana
  - Canton, Ohio
  - Portland, Oregon
  - Greer, South Carolina
  - Midland, Texas
  - Richmond, Virginia
- Estonia (2):
  - Tallinn
  - Tartu
- Latvia (2):
  - Jelgava
  - Riga
- Mexico (3):
  - Chihuahua City
  - Guadalajara
  - Pachuca